CLINICAL TRIAL: NCT02980172
Title: Pain Evaluation and Treatment in the Emergency Department
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Olivier T. Rutschmann, Professor, Deputy Chief, University Hospital, Geneva
Other Study IDs: CCER 2016-00205
Record Dates: First submitted 2016-11-24; First posted 2016-12-02 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Pain, Acute; Emergencies
Keywords: triage
MeSH Terms: conditions — Acute Pain; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pain triage complaint: Patients admitted at GUH ED triaged with a main complaint requiring a pain evaluation.
  Interventions: Other: Pain evaluation

INTERVENTIONS:
Other: Pain evaluation — Evaluation of pain using a numerical scale (1 to 10)

SUMMARY:
All patients admitted in Geneva University Hospitals (GUH) emergency department (ED) are triaged using the Swiss Emergency Triage Scale (SETS), a 4-level symptom-based triage scale. At the end of the triage process the triage nurse has to choose an emergency level and a main presenting complaint among a listing of 98 presenting complaints. The SETS recommends a pain evaluation for 44 out of the SETS 98 presenting complaint.

The primary objective of the study is to determine whether pain is correctly evaluated when required by the SETS criteria. The secondary objectives are (1) to evaluate whether an appropriate treatment is delivered when pain is present, and (2) to identify predictors of pain evaluation and treatment.

DETAILED DESCRIPTION:
All patients admitted in Geneva University Hospitals (GUH) emergency department (ED) are triaged using the Swiss Emergency Triage Scale (SETS), a 4-level symptom-based triage scale. At the end of the triage process the triage nurse has to choose an emergency level and a main presenting complaint among a listing of 98 presenting complaints. The SETS recommends a pain evaluation for 44 out of the SETS 98 presenting complaint.

After this evaluation, a protocol standardize administration of analgesia for patients presenting pain.

The primary objective of the study is to determine whether pain is correctly evaluated when required by the SETS criteria for the 44 presenting complaints.

The secondary objectives are (1) to evaluate whether an appropriate treatment is delivered when pain is present, and (2) to identify predictors of pain evaluation and treatment.

ELIGIBILITY:
Inclusion Criteria:

* adult (>= 16y) patients admitted at GUH ED during one year
* presenting complaint requiring pain evaluation accordingly to the SETS criteria

Exclusion Criteria:

* < 16 y
* presenting complaint that does not require a pain evaluation accordingly to the SETS criteria

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted during one year at GUH ED.
Sampling Method: Non-Probability Sample
Enrollment: 31942 (Actual)
Dates: Start 2016-11; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with appropriate pain evaluation | Within 24 hours after ED admission
  Percentage of patients with a documented assessement of pain using a numerical scale (0 to 10)

SECONDARY OUTCOMES:
Proportion of patients with appropriate pain treatment | Within 24 hours after ED admission
  Percentage of patients who received an appropriate treatment accordingly to the ED recommendations.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier T Rutschmann, MD, MPH, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals, ED, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No